CLINICAL TRIAL: NCT03607019
Title: Epidemiology and Prognostic Impact of Social Deprivation Features in Intensive Care Unit Patients
Brief Title: Social Deprivation Features in Intensive Care Unit Patients
Acronym: PRECAREA
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier de Saint-Denis (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-A01272-51
Record Dates: First submitted 2018-07-13; First posted 2018-07-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-03

CONDITIONS: Socioeconomic Factors
Keywords: Intensive care; Critical care; Poverty; inequalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Socioeconomic inequalities are increasingly recognised as an important public health issue, and it is now well established that patients with socioeconomic deprivation (SED) features demonstrate higher mortality and morbidity. The epidemiology and impact of SED on the specific population of ICU patients has been insufficiently investigated.

In this prospective multicenter study of patients admitted to 9 ICUs of the Paris area, the investigators aim to explore the epidemiology of SED features, and its impact on mortality and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admission to one of the participating intensive care units

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted to one of the participating ICUs during the study period
Sampling Method: Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-09-15 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
30-day mortality | 30 days
  30-day mortality

SECONDARY OUTCOMES:
ICU length of stay | up to 12 weeks
  ICU length of stay
Hospital length of stay | up to 12 weeks
  Hospital length of stay
ICU mortality | up to 12 weeks
  ICU mortality

OTHER OUTCOMES:
30-day mortality of pre-specified subgroup of undocumented immigrants | 30 days
  30-day mortality of pre-specified subgroup of patients who are undocumented
30-day mortality of pre-specified subgroup of deprived patients aged between 18 and 25 years old | 30 days
  30-day mortality of pre-specified subgroup of deprived patients (ie without healthcare coverage and/or without income and/or without housing) aged between 18 and 25 years old

CONTACTS AND LOCATIONS:
Overall Officials: Etienne de Montmollin, MD, Principal Investigator — Centre Hospitalier de Saint-Denis; Morgan Benais, MD, Study Chair — Centre Hospitalier de Saint-Denis; Daniel Da Silva, MD, Study Chair — Centre Hospitalier de Saint-Denis
Locations (9):
- France (9):
  - Centre Hospitalier Universitaire Ambroise Paré, Boulogne-Billancourt
  - Centre Hospitalier Universitaire Louis Mourier, Colombes
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Grand Hopital de l'Est Francilien, Jossigny
  - Groupe Hospitalier Nord-Essone, Longjumeau
  - Centre Hospitalier Intercommunal André Grégoire, Montreuil
  - Centre Hospitalier Universitaire Lariboisière, Paris
  - Centre Hospitalier de Saint-Denis, Saint-Denis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marmot M, Allen J, Bell R, Bloomer E, Goldblatt P; Consortium for the European Review of Social Determinants of Health and the Health Divide. WHO European review of social determinants of health and the health divide. Lancet. 2012 Sep 15;380(9846):1011-29. doi: 10.1016/S0140-6736(12)61228-8. Epub 2012 Sep 8. PMID 22964159
- [Background] Welch CA, Harrison DA, Hutchings A, Rowan K. The association between deprivation and hospital mortality for admissions to critical care units in England. J Crit Care. 2010 Sep;25(3):382-90. doi: 10.1016/j.jcrc.2009.11.003. Epub 2010 Jan 15. PMID 20074907
- [Background] Zager S, Mendu ML, Chang D, Bazick HS, Braun AB, Gibbons FK, Christopher KB. Neighborhood poverty rate and mortality in patients receiving critical care in the academic medical center setting. Chest. 2011 Jun;139(6):1368-1379. doi: 10.1378/chest.10-2594. Epub 2011 Mar 31. PMID 21454401
- [Background] Latour J, Lopez V, Rodriguez M, Nolasco A, Alvarez-Dardet C. Inequalities in health in intensive care patients. J Clin Epidemiol. 1991;44(9):889-94. doi: 10.1016/0895-4356(91)90051-a. PMID 1890431
- [Background] Bein T, Hackner K, Zou T, Schultes S, Bosch T, Schlitt HJ, Graf BM, Olden M, Leitzmann M. Socioeconomic status, severity of disease and level of family members' care in adult surgical intensive care patients: the prospective ECSSTASI study. Intensive Care Med. 2012 Apr;38(4):612-9. doi: 10.1007/s00134-012-2463-x. Epub 2012 Jan 25. PMID 22273749
- [Background] Bige N, Hejblum G, Baudel JL, Carron A, Chevalier S, Pichereau C, Maury E, Guidet B. Homeless Patients in the ICU: An Observational Propensity-Matched Cohort Study. Crit Care Med. 2015 Jun;43(6):1246-54. doi: 10.1097/CCM.0000000000000944. PMID 25793435